CLINICAL TRIAL: NCT05459051
Title: Finding the Invasive Haemodynamic Threshold for Symptom Relief in Stable Angina
Acronym: ORBITA-FIRE
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: P91528; 22HH7546 (Other: Imperial College London)
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Stable Angina
Keywords: Symptoms; Angina; Physiology; Placebo
MeSH Terms: conditions — Angina, Stable; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stable angina: * Symptomatic
  * Anatomically severe single-vessel coronary artery disease
  * Physiological evidence of myocardial ischaemia
  Interventions: Diagnostic Test: Rest-angina physiological assessment; Diagnostic Test: Exercise-angina physiological assessment

INTERVENTIONS:
Diagnostic Test: Rest-angina physiological assessment — The degree of stenosis required to cause angina at rest will be measured under double-blinded placebo controlled conditions using sequential intracoronary balloon inflations. This will then be correlated with various physiological indices, including FFR and NHPR.
Diagnostic Test: Exercise-angina physiological assessment — The degree of stenosis required to cause angina during exercise will be measured under double-blinded placebo controlled conditions using sequential intracoronary balloon inflations. This will then be correlated with various physiological indices, including FFR and NHPR.

SUMMARY:
ORBITA-FIRE is a randomised, double-blinded, placebo controlled experimental study that will identify the fractional flow reserve (FFR) and non-hyperemic pressure ratio (NHPR) thresholds that correlate with symptoms of angina for 58 patients measured invasively under experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for percutaneous coronary intervention (PCI) due to angina or angina-equivalent symptoms on exertion
* Anatomical evidence of significant single-vessel coronary stenosis defined by either:

  * ≥70% stenosis on invasive coronary angiography (ICA)
  * Severe stenosis on CT coronary angiography (CTCA)
* Physiological evidence of ischaemia with a positive test on at least one of the following:

  * Stress echocardiography
  * Cardiac magnetic resonance perfusion
  * Myocardial perfusion scintigraphy
  * Invasive metrics of coronary physiology

Exclusion Criteria:

* Age <18 years
* Recent acute coronary syndrome
* Previous coronary artery by-pass graft
* Significant left main stem disease
* Multivessel disease (defined as >50% angiographic stenosis in other vessels)
* Chronic total occlusion in the target artery
* Moderate to severe valvular disease
* Moderate to severe left ventricular impairment
* Chronotropic incompetence with a pacemaker
* Contraindication to PCI or a drug-eluting stents
* Contraindication to antiplatelet therapy
* Contraindication to adenosine
* Moderate to severe respiratory disease
* Physical inability to exercise
* Pregnant
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with stable angina
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
The FFR and NHPR value at which the patient experiences angina in a rest state | Intra-procedural
  Values 0.00-1.00 (Lower = More significant disease)
The FFR and NHPR value at which the patient experiences angina in an exercise state | Intra-procedural
  Values 0.00-1.00 (Lower = More significant disease)

SECONDARY OUTCOMES:
The FFR difference between the rest and exercise states | Intra-procedural
  Values 0.00-1.00 (Lower = More significant disease)
The NHPR difference between the rest and exercise states | Intra-procedural
  Values 0.00-1.00 (Lower = More significant disease)
Angina severity score at the angina threshold | Intra-procedural
  The patient scores the severity of the angina experienced during the procedure between 0-10 (Higher = More severe)
Angina similarity score at the angina threshold | Intra-procedural
  The patient scores the similarity of the angina experienced during the procedure against the angina experienced before the procedure between 0-10 (Higher = Most similar)
Angina symptom type at the angina threshold | Intra-procedural
  The patient will list all symptoms experienced at the angina threshold

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Al-Lamee, PhD MRCP, Principal Investigator — Imperial College London
Locations (6):
- United Kingdom (6):
  - Mid and South Essex NHS Foundation Trust, Basildon
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Imperial College NHS Trust, London
  - Royal Free Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No